CLINICAL TRIAL: NCT04660539
Title: A Multicenter, Single Arm, Open-Label Study to Evaluate the Long-Term Safety and Efficacy of Satralizumab in Patients With Neuromyelitis Optica Spectrum Disorder (NMOSD)
Brief Title: A Study to Evaluate the Safety and Efficacy of Satralizumab in Participants With Neuromyelitis Optica Spectrum Disorder (NMOSD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WN42349; 2020-003413-35 (EudraCT Number)
Record Dates: First submitted 2020-11-24; First posted 2020-12-09 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-11

CONDITIONS: Neuromyelitis Optica Spectrum Disorder
MeSH Terms: conditions — Neuromyelitis Optica | interventions — satralizumab; Azathioprine; Mycophenolic Acid; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Satralizumab Treatment (Experimental): Participants will receive satralizumab subcutaneously (SC) every 4 weeks (Q4W)
  Interventions: Drug: satralizumab; Drug: azathioprine (AZA); Drug: mycophenolate mofetil (MMF); Drug: oral corticosteroids

INTERVENTIONS:
Drug: satralizumab — Satralizumab will be administered by SC injection in the abdominal or femoral region at a dose of 120 mg (fixed dose) Q4W for up to 3 years
  Other Names: Enspryng
Drug: azathioprine (AZA) — Participants are permitted to use AZA during the study as background immunosuppressive treatment at a maximum dose of 3 milligram per kilogram per day (mg/kg/day)
  Other Names: non-investigational medicinal product (NIMP)
Drug: mycophenolate mofetil (MMF) — Participants are permitted to use MMF during the study as background immunosuppressive treatment at a maximum dose of 3000 mg/day
  Other Names: NIMP
Drug: oral corticosteroids — Participants are permitted to use oral corticosteroids (prednisolone equivalent) during the study as background immunosuppressive treatment at a maximum dose of 15 mg/day
  Other Names: NIMP

SUMMARY:
This multicenter, single-arm, open-label study will evaluate the long-term safety and efficacy of satralizumab in participants with neuromyelitis optica spectrum disorder (NMOSD) who completed open-label extension (OLE) period of studies BN40898 and BN40900. Participants will receive satralizumab as monotherapy or in combination with one of the following background immunosuppressive treatments: azathioprine (AZA), mycophenolate mofetil (MMF), or oral corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged less than 18 years at the time of informed consent for Study BN40898 can continue treatment with a combination of oral corticosteroids and either AZA or MMF
* Participated in Study BN40898 or Study BN40900 with satralizumab in NMOSD, are on ongoing satralizumab treatment and were anti-aquaporin-4 IgG antibody (AQP4-IgG) seropositive at screening in these studies. Participants with NMOSD who were AQP4-IgG seronegative at screening in Study BN40898 or Study BN40900 can be enrolled if the investigator considers the continued treatment with satralizumab to be beneficial for the participant
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use adequate contraception during the treatment period and for 3 months after the final dose of satralizumab.

Exclusion Criteria:

* Pregnant or breastfeeding, or intending to become pregnant during the study or within 3 months after the final dose of study drug. Women of childbearing potential must have a negative urine pregnancy test result on the baseline visit prior to initiation of study drug
* Evidence of any serious uncontrolled concomitant diseases that may preclude participation including nervous system disease, cardiovascular disease, hematologic/hematopoiesis disease, respiratory disease, muscular disease, endocrine disease, renal/urologic disease, digestive system disease, congenital or acquired severe immunodeficiency
* Known active infection that requires delaying the next satralizumab dose at the time of enrollment
* NMOSD relapse at the time of enrollment
* Laboratory abnormalities at the last assessment in Study BN40898 or Study BN40900 that preclude re-treatment with satralizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (53):
- United States (13):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Miami, Miami, Florida
  - Columbus Research and Wellness, Columbus, Georgia
  - University of Chicago, Chicago, Illinois
  - Consultants in Neurology Ltd, Northbrook, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Wayne State University; UHC-4H, Detroit, Michigan
  - The Neurological Institute PA, Charlotte, North Carolina
  - OhioHealth Research Institute, Columbus, Ohio
  - Jefferson Hospital For Neuroscience; Jefferson Neurology Associates, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
- Bulgaria (3):
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - Multiprofile Hospital for Active Treatment of Neurology and Psychiatry Sv. Naum EAD, Sofia
  - University Multiprofile Hospital for Active Treatment Aleksandrovska EAD, Sofia
- Canada (2):
  - MS Clinical Trials Group, Vancouver, British Columbia
  - Centre hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
- Clinical Hospital Centre Osijek, Osijek, Croatia
- Ruhr Universitat Bochum, Bochum, Germany
- Jahn Ferenc Del-Pesti Korhaz es Rendelointezet, Budapest, Hungary
- Italy (2):
  - Azienda Ospedaliera Sant'Andrea, Rome, Lazio
  - Azienda Ospedaliero Universitaria Policlinico Vittorio Emanuele, Catania, Sicily
- Japan (7):
  - Kyushu University Hospital, Fukuoka
  - Tohoku University Hospital, Miyagi
  - Niigata University Medical & Dental Hospital, Niigata
  - Osaka University Hospital, Osaka
  - Kindai University Hospital, Osaka
  - Tokyo Women's Medical University Hospital, Tokyo
  - National Center of Neurology and Psychiatry, Tokyo
- Hospital Kuala Lumpur, Kuala Lumpur, FED. Territory of Kuala Lumpur, Malaysia
- Poland (6):
  - NZOZ Wielospecjalistyczna Poradnia Lekarska SYNAPSIS, Katowice
  - M.A. - LEK A. M. Maciejowscy SC. Centrum Terapii SM, Katowice
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie; Klinika Neurologii, Lublin
  - Uniwersyteckie Centrum Kliniczne WUM, Centralny Szpital Kliniczny; Klinika Neurologii, Warsaw
  - Instytut Psychiatrii i Neurologii, Warsaw
  - Miedzyleski Szpital Specjalistyczny w Warszawie, Warsaw
- San Juan MS Center, Guaynabo, Puerto Rico
- SC Clubul Sanatatii SRL, Campulung Muscel, Romania
- South Korea (2):
  - Korea University Anam Hospital, Seoul
  - Asan Medical Center - PPDS, Seoul
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona
  - Hosp. Clinico San Carlos, Madrid
- Taiwan (4):
  - China Medical University Hospital, North Dist.
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Bilim University Medical Faculty Florence Nightingale Hospital, Istanbul, Turkey (Türkiye)
- Ukraine (4):
  - Municipal Non-Profit Enterprise City Clinical Hospital #16 of Dnipro City Council, Dnipro, Katerynoslav Governorate
  - Municipal Non-Commercial Enterprise Odesa RMC for Mental Health of Odessa Regional Council, Odesa, Kherson Governorate
  - Communal NPE Vinnytsia Reg. Clin. Psychoneurolog. Hosp. n.a. O.I. Yushchenko of Vinnytsia RC, Vinnytsia, Podolia Governorate
  - Communal Nonprofit enterprise Ternopil Regional Clinical Psychoneurological Hospital of TRC, Ternopil, Volhynian Governorate
- National Hospital For Neurology and Neurosurgery, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Bennett JL, Fujihara K, Saiz A, Traboulsee AL, Greenberg BM, Weinshenker BG, Patti F, Kleiter I, Palace J, De Seze J, Evans R, Blondeau K, Klingelschmitt G, Vodopivec I, Rahim M, Yamamura T. Long-Term Efficacy and Safety of Satralizumab in Patients With Neuromyelitis Optica Spectrum Disorder From the SAkuraMoon Open-Label Extension Study. Neurol Neuroimmunol Neuroinflamm. 2025 Sep;12(5):e200450. doi: 10.1212/NXI.0000000000200450. Epub 2025 Jul 31. PMID 40743487

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 119 participants with neuromyelitis optica spectrum disorder (NMOSD) who completed open-label extension (OLE) period of studies BN40898 (NCT02028884) & BN40900 (NCT02073279) rolled over in study WN42349 at 53 sites in 17 countries. 'All Participants-treated population' is used to report results of this study, which includes 166 participants who received at least one dose of satralizumab at any time either during parent studies/this study, irrespective of enrollment in current study.
Pre-assignment Details: Participants from NCT02028884 and NCT02073279 enrolled in this study to receive satralizumab treatment. Participants were permitted to use azathioprine (AZA) or mycophenolate mofetil (MMF) or oral corticosteroids during the study as background immunosuppressive treatments.
Groups:
- Satralizumab: Participants rolled over from studies NCT02028884 and NCT02073279 received satralizumab, 120 milligrams (mg) as subcutaneous (SC) injection, every 4 weeks (Q4W) up to a maximum duration of 3 years in this study. Participants who received at least 1 dose of satralizumab at any time during the parent studies or this study, irrespective of enrollment in current study are represented here.
Period: Overall Study
Arm/Group | Satralizumab
Started | 166
Completed | 106
Not Completed | 60
Not completed — Adverse Event | 10
Not completed — Lack of Efficacy | 4
Not completed — Lost to Follow-up | 5
Not completed — Non-Compliance With Study Drug | 3
Not completed — Reason not Specified | 12
Not completed — Pregnancy | 2
Not completed — Protocol Violation | 2
Not completed — Switch To Commercial Satralizumab | 1
Not completed — Withdrawal by Subject | 21

BASELINE CHARACTERISTICS:
Population: All Participants-treated population included all participants who received at least one dose of satralizumab at any time either during the parent studies or this study.
Groups:
- Satralizumab: Participants rolled over from studies NCT02028884 and NCT02073279 received satralizumab, 120 mg as SC injection, Q4W up to a maximum duration of 3 years in this study. Participants who received at least 1 dose of satralizumab at any time during the parent studies or this study, irrespective of enrollment in current study are represented here.
Arm/Group | Satralizumab
Number analyzed (Participants) | 166
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 147
  Unknown or Not Reported | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 47
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 95
  More than one race | 0
  Other | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE=any untoward medical occurrence in a participant administered a pharmaceutical product, regardless of causal relationship with it. AE can therefore be any unfavorable & unintended sign, symptoms/disease temporally associated with use of a medicinal (investigational) product, whether or not considered related to it. SAE is any significant hazard, contraindication, or side effect that is fatal or life-threatening, requires hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is medically significant or requires intervention. The first dosing visit in the current study or randomization visit in the parent studies (NCT02028884/NCT02073279) was considered as baseline for this outcome measure. All AEs from the time of randomization in the parent studies for satralizumab-treated participants are reported here.
Time Frame: Baseline up to 523 weeks
Population: All Participants-treated population included participants who received at least one dose of satralizumab at any time either during the parent studies or this study, irrespective of enrollment in current study.
Measure: Count of Participants; unit: Participants
Arm/Group | Satralizumab
Number analyzed (Participants) | 166
Participants
  AEs | 162
  SAEs | 44

2. Primary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs) and Selected AEs
Description: An AESIs included potential drug induced liver injury and suspected transmission of an infectious agent by study drug defined as any organism, virus, or infectious particle (e.g., prion protein transmitting transmissible spongiform encephalopathy), pathogenic or non-pathogenic causing clinical symptoms or laboratory findings that indicate an infection in a participant exposed to a medicinal product. Selected AEs included infections that required treatments with IV antibiotics, antifungals, or antivirals; opportunistic infections that required treatment with oral antibiotics, antifungals, or antivirals and injection related reaction. The first dosing visit in the current study or randomization visit in the parent studies (NCT02028884/NCT02073279) was considered as baseline for this outcome measure. All AEs from the time of randomization in the parent studies for satralizumab-treated participants are reported here.
Time Frame: Baseline up to 523 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Satralizumab
Number analyzed (Participants) | 166
Participants
  AESIs | 0
  Selected AEs | 0

3. Secondary Outcome: Number of Participants With Suicidality Assessed Using Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS=assessment tool used to assess lifetime suicidality of a participant (at baseline) as well as any new instances of suicidality (since last visit). Structured interview prompts recollection of suicidal ideation, including intensity of ideation, behavior & attempts with actual/potential lethality. Categories have binary responses (yes/no) & include a-Wish to be Dead; b-Non-specific Active Suicidal Thoughts; c-Active Suicidal Ideation with Any Methods(Not Plan) without Intent to Act; d-Active Suicidal Ideation with Some Intent to Act, without Specific Plan; e-Active Suicidal Ideation with Specific Plan & Intent, f-Preparatory Acts & Behavior; g-Aborted Attempt; h-Interrupted Attempt; i-Actual Attempt(non-fatal); j-Completed Suicide. Suicidal ideation/behavior is indicated by a "yes" answer to any of listed categories. Score of 0 is assigned if no suicide risk is present. Score of 1 or higher= suicidal ideation or behavior. Categories with non-zero values are only reported here.
Time Frame: Baseline up to 523 weeks
Population: All Participants-treated population included participants who received at least one dose of satralizumab at any time either during the parent studies or this study. The first dosing visit in the current study or randomization visit in the parent studies (NCT02028884/NCT02073279) was considered as baseline for this outcome measure. All data from the time of randomization in the parent studies for satralizumab-treated participants are reported here.
Measure: Count of Participants; unit: Participants
Arm/Group | Satralizumab
Number analyzed (Participants) | 166
Participants
  a- Baseline | 7
  a- Post-baseline | 5
  b- Baseline | 5
  b- Post-baseline | 2
  c- Baseline | 1
  c- Post-baseline | 0
  d- Baseline | 1
  d- Post-baseline | 0
  e- Baseline | 1
  e- Post-baseline | 0
  f- Baseline | 2
  f- Post-baseline | 0
  i- Baseline | 3
  i- Post-baseline | 1
  j- Baseline | 0
  j- Post-baseline | 1

4. Secondary Outcome: Number of Participants With Serious Infections and Hepatotoxicity
Description: Hepatotoxicity was defined using the following Medical Dictionary for Regulatory Activities Standardised MedDRA Queries (MedDRA SMQs) - Cholestasis and jaundice of hepatic origin (SMQ narrow) and Drug related hepatic disorders - severe events only (SMQ narrow). The first dosing visit in the current study or randomization visit in the parent studies (NCT02028884/NCT02073279 ) was considered as baseline for this outcome measure. Data for all serious infections and hepatotoxicity from the time of randomization in the parent studies for satralizumab-treated participants are reported here.
Time Frame: Baseline up to 523 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Satralizumab
Number analyzed (Participants) | 166
Participants
  Serious Infections | 19
  Hepatotoxicity | 8

5. Secondary Outcome: Time to First Protocol-defined Relapse (PDR) as Assessed by Investigator (iPDR)
Description: Time to first relapse (TFR) was defined as the time from randomization in parent studies to the first occurrence of the first iPDR. PDR=occurrence of new or worsening neurological symptoms attributable to neurological neuromyelitis optica (NMO) or NMOSD. New or worsening neurological symptoms that occur < 31 days following onset of PDR were considered part of same relapse. The time point of relapse onset=time at which the participant experienced any new or worsening neurological symptoms representing NMOSD clinical relapse(s). For participants who did not relapse at the time of analysis, TFR was censored at the clinical cutoff date (CCOD) or at the time of withdrawal from study. The first dosing visit in current study or randomization visit in the parent studies (NCT02028884/NCT02073279) was considered as baseline. All TFR data from the time of randomization in the parent studies up to the end of study WN42349 for satralizumab-treated participants are reported here.
Time Frame: Baseline up to 528 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Satralizumab
Number analyzed (Participants) | 166
weeks | NA [NA to NA] — Median and 95% CI was not estimable because there was an insufficient number of participants with events.

6. Secondary Outcome: iPDR-free Rate up to Week 456
Description: iPDR free rate was defined as the percentage of participants who did not experience a protocol-defined relapse as assessed by the investigator. Protocol-defined relapse was the occurrence of new or worsening neurological symptoms attributable to NMOSD. New or worsening neurological symptoms that occur < 31 days following the onset of a PDR were considered part of the same relapse. The first dosing visit in the current study or randomization visit in the parent studies (NCT02028884/NCT0207327) was considered as baseline for this outcome measure. All data from the time of randomization in the parent studies up to Week 456 for satralizumab-treated participants are reported here. Percentages have been rounded off to the nearest decimal point. Kaplan-Meier method was used to estimate the iPDR-free rates.
Time Frame: Baseline up to Week 456
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Satralizumab
Number analyzed (Participants) | 166
percentage of participants | 67.11 [58.61 to 74.25]

7. Secondary Outcome: Percentage of Relapse-Free Participants
Description: Protocol-defined relapse was the occurrence of new or worsening neurological symptoms attributable to NMOSD. New or worsening neurological symptoms that occur < 31 days following the onset of a PDR were considered part of the same relapse. The first dosing visit in the current study or randomization visit in the parent studies (NCT02028884/NCT0207327) was considered as baseline for this outcome measure. All data from the time of randomization in the parent studies up to end of study WN42349 for satralizumab-treated participants are reported here. Participants who did not experience any relapse events are reported here. Percentages have been rounded off to the nearest decimal point.
Time Frame: Baseline up to 528 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Satralizumab
Number analyzed (Participants) | 166
percentage of participants | 70.5 [58.61 to 74.25]

8. Secondary Outcome: Annualized Relapse Rate (ARR)
Description: ARR was calculated as total number of relapses experienced divided by the participant-years of the whole study period. Adjusted ARR was calculated using Poisson regression model adjusted by study identifier (BN40898, BN40900). ARR was assessed from randomization in parent studies to the first occurrence of the iPDR. PDR=occurrence of new/worsening neurological symptoms attributable to NMO/NMOSD. New or worsening neurological symptoms that occur < 31 days following onset of a PDR were considered part of the same relapse. Time point of relapse onset=the time at which the participant experienced any new or worsening neurological symptoms representing NMOSD clinical relapse(s). First dosing visit in the current study or randomization visit in the parent studies (NCT02028884/NCT02073279) was considered as baseline for this outcome measure. All ARR data from time of randomization in the parent studies up to the end of study WN42349 for satralizumab-treated participants are reported here.
Time Frame: Baseline up to 528 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: relapses per participant-year
Arm/Group | Satralizumab
Number analyzed (Participants) | 166
relapses per participant-year | 0.0788 [0.0633 to 0.0982]

9. Secondary Outcome: Change in Expanded Disability Status Scale (EDSS) Score
Description: EDSS was a quantitative measure of disability and for assessment of severity of relapse for participants with NMOSD. Values from 0 points (normal neurological examination) up to 10 points (death), increasing in increments of 0.5 points. Higher scores represent increased disability. Baseline is the last observation on or before the day of first study drug administration in the current study or the parent studies (NCT02028884/NCT02073279). All EDSS data from the time of randomization in the parent studies up to the end of study WN42349 for satralizumab-treated participants are reported here.
Time Frame: Baseline and every 24 weeks (up to 528 weeks)
Population: All Participants-treated population included participants who received at least one dose of satralizumab at any time either during the parent studies or this study, irrespective of enrollment in the current study. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Satralizumab
Number analyzed (Participants) | 165
score on a scale
  Baseline | 3.80 (1.57)
  Change from Baseline at Week 24: number analyzed (Participants) | 162
  Change from Baseline at Week 24 | -0.08 (0.77)
  Change from Baseline at Week 48: number analyzed (Participants) | 151
  Change from Baseline at Week 48 | -0.16 (0.72)
  Change from Baseline at Week 72: number analyzed (Participants) | 147
  Change from Baseline at Week 72 | -0.14 (0.80)
  Change from Baseline at Week 96: number analyzed (Participants) | 141
  Change from Baseline at Week 96 | -0.18 (0.86)
  Change from Baseline at Week 120: number analyzed (Participants) | 135
  Change from Baseline at Week 120 | -0.14 (0.90)
  Change from Baseline at Week 144: number analyzed (Participants) | 133
  Change from Baseline at Week 144 | -0.09 (0.97)
  Change from Baseline at Week 168: number analyzed (Participants) | 128
  Change from Baseline at Week 168 | -0.16 (0.90)
  Change from Baseline at Week 192: number analyzed (Participants) | 129
  Change from Baseline at Week 192 | -0.13 (0.95)
  Change from Baseline at Week 216: number analyzed (Participants) | 124
  Change from Baseline at Week 216 | -0.22 (0.99)
  Change from Baseline at Week 240: number analyzed (Participants) | 116
  Change from Baseline at Week 240 | -0.21 (0.95)
  Change from Baseline at Week 264: number analyzed (Participants) | 114
  Change from Baseline at Week 264 | -0.25 (0.92)
  Change from Baseline at Week 288: number analyzed (Participants) | 106
  Change from Baseline at Week 288 | -0.34 (0.99)
  Change from Baseline at Week 312: number analyzed (Participants) | 97
  Change from Baseline at Week 312 | -0.44 (1.02)
  Change from Baseline at Week 336: number analyzed (Participants) | 87
  Change from Baseline at Week 336 | -0.42 (1.15)
  Change from Baseline at Week 360: number analyzed (Participants) | 82
  Change from Baseline at Week 360 | -0.51 (1.24)
  Change from Baseline at Week 384: number analyzed (Participants) | 66
  Change from Baseline at Week 384 | -0.37 (1.22)
  Change from Baseline at Week 408: number analyzed (Participants) | 52
  Change from Baseline at Week 408 | -0.26 (1.20)
  Change from Baseline at Week 432: number analyzed (Participants) | 48
  Change from Baseline at Week 432 | -0.31 (1.16)
  Change from Baseline at Week 456: number analyzed (Participants) | 37
  Change from Baseline at Week 456 | -0.31 (1.23)
  Change from Baseline at Week 480: number analyzed (Participants) | 16
  Change from Baseline at Week 480 | 0.00 (1.03)
  Change from Baseline at Week 504: number analyzed (Participants) | 1
  Change from Baseline at Week 504 | 0.00 (NA) — Since only 1 participant was analyzed, standard deviation (SD) could not be calculated.
  Change from Baseline at Week 528: number analyzed (Participants) | 1
  Change from Baseline at Week 528 | -0.50 (NA) — Since only 1 participant was analyzed, SD could not be calculated.

10. Secondary Outcome: Time to First EDSS Scores Worsening
Description: EDSS=quantitative measure of disability & for assessment of severity of relapse for participants with NMOSD. Values from 0 points (normal neurological examination) up to 10 points (death), increasing in increments of 0.5 points. Higher scores=increased disability. EDSS worsening=(a) worsening of 2/more points in EDSS score for participants with a baseline score (BS) of 0, (b) worsening of 1/more points in EDSS score for participants with a BS of 1 to 5, or (c) worsening of 0.5 points/more in EDSS score for participants with a BS of 5.5/more. Participants were censored at date of last EDSS assessment or if no EDSS assessment was performed at randomization date. Baseline=last observation on/before day of first study drug administration in current study/parent studies (NCT02028884/NCT02073279). All EDSS data from time of randomization in parent studies up to end of study WN42349 for satralizumab-treated participants are reported here.
Time Frame: Baseline up to 528 weeks
Population: All Participants-treated population included participants who received at least one dose of satralizumab at any time either during the parent studies or this study, irrespective of enrollment in the current study. Overall number analyzed is the number of participants with data available for analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Satralizumab
Number analyzed (Participants) | 165
weeks | NA [398.1 to NA] — Median and upper limit of 95% CI was not estimable because there was an insufficient number of participants with events.

11. Secondary Outcome: Event-free Rate for EDSS Score Worsening up to Week 456
Description: Event-free rate for EDSS score worsening was defined as the percentage of participants who did not experience worsening in their EDSS score from baseline. EDSS=quantitative measure of disability & for assessment of severity of relapse for participants with NMOSD. Values from 0 points (normal neurological examination) up to 10 points (death), increasing in increments of 0.5 points. Higher scores=increased disability. Participants were censored at the date of the last EDSS assessment or if no EDSS assessment was performed at the randomization date. Baseline is defined as the last observation on/before the day of the first study drug administration in current study/parent studies (NCT02028884/NCT02073279). All EDSS data from the time of randomization in the parent studies up to Week 456 for satralizumab-treated participants are reported here. Kaplan-Meier method was used to estimate the event-free rates.
Time Frame: Baseline up to Week 456
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Satralizumab
Number analyzed (Participants) | 165
percentage of participants | 57.03 [46.80 to 66.01]

12. Secondary Outcome: Percentage of Participants Without EDSS Worsening
Description: EDSS=quantitative measure of disability & for assessment of severity of relapse for participants with NMOSD. Values from 0 points (normal neurological examination) up to 10 points (death), increasing in increments of 0.5 points. Higher scores=increased disability. EDSS worsening=(a) worsening of 2/more points in EDSS score for participants with a BS of 0, (b) worsening of 1/more points in EDSS score for participants with a BS of 1 to 5, or (c) worsening of 0.5 points/more in EDSS score for participants with a BS of 5.5/more. Baseline=last observation on/before day of first study drug administration in current study/parent studies (NCT02028884/NCT02073279). All EDSS data from time of randomization in parent studies up to end of study WN42349 for satralizumab-treated participants are reported here. Participants who did not experience any EDDS worsening events are reported here. Percentages have been rounded off to the nearest decimal point.
Time Frame: Baseline up to 528 weeks
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Satralizumab
Number analyzed (Participants) | 165
percentage of participants | 64.8

13. Secondary Outcome: Change in Visual Acuity (VA) Assessed by a Snellen 20-Foot Wall Chart
Description: Visual acuity is measured using Snellen 20-foot wall chart and then converted to logMAR visual acuity scoring. Lower values indicate better visual acuity. Data are reported for right eye (OD) and left eye (OS). Visual acuity scores (Snellen chart) worse than 20/200 [i.e. CF (counting fingers), HM (hand movement), LP (light perception), or NLP (no LP)] are converted to logMAR 1.85, logMAR 2.00, logMAR 2.70, and logMAR 3.00 respectively. LogMAR >= 1 is equivalent to Physically blind. A negative change from baseline indicates an improvement. The first dosing visit in the current study or randomization visit in the parent studies (NCT02028884/NCT02073279) was considered as baseline for this outcome measure. All VA data from the time of randomization in the parent studies up to the end of study WN42349 for satralizumab-treated participants are reported here.
Time Frame: Baseline and every 24 weeks (up to 528 weeks)
Population: All Participants-treated population included participants who received at least one dose of satralizumab at any time either during the parent studies or this study, irrespective of enrollment in the current study. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: LogMAR units
Arm/Group | Satralizumab
Number analyzed (Participants) | 166
LogMAR units
  Baseline [OD] | 0.438 (0.746)
  Baseline [OS] | 0.566 (0.899)
  Change from Baseline at Week 24 [OD]: number analyzed (Participants) | 162
  Change from Baseline at Week 24 [OD] | 0.028 (0.297)
  Change from Baseline at Week 24 [OS]: number analyzed (Participants) | 161
  Change from Baseline at Week 24 [OS] | 0.009 (0.329)
  Change from Baseline at Week 48 [OD]: number analyzed (Participants) | 152
  Change from Baseline at Week 48 [OD] | 0.014 (0.363)
  Change from Baseline at Week 48 [OS]: number analyzed (Participants) | 152
  Change from Baseline at Week 48 [OS] | 0.020 (0.385)
  Change from Baseline at Week 72 [OD]: number analyzed (Participants) | 148
  Change from Baseline at Week 72 [OD] | -0.004 (0.340)
  Change from Baseline at Week 72 [OS]: number analyzed (Participants) | 147
  Change from Baseline at Week 72 [OS] | -0.017 (0.362)
  Change from Baseline at Week 96 [OD]: number analyzed (Participants) | 141
  Change from Baseline at Week 96 [OD] | -0.024 (0.375)
  Change from Baseline at Week 96 [OS]: number analyzed (Participants) | 141
  Change from Baseline at Week 96 [OS] | -0.030 (0.317)
  Change from Baseline at Week 120 [OD]: number analyzed (Participants) | 136
  Change from Baseline at Week 120 [OD] | 0.015 (0.404)
  Change from Baseline at Week 120 [OS]: number analyzed (Participants) | 135
  Change from Baseline at Week 120 [OS] | -0.065 (0.404)
  Change from Baseline at Week 144 [OD]: number analyzed (Participants) | 134
  Change from Baseline at Week 144 [OD] | -0.023 (0.379)
  Change from Baseline at Week 144 [OS]: number analyzed (Participants) | 134
  Change from Baseline at Week 144 [OS] | -0.054 (0.355)
  Change from Baseline at Week 168 [OD]: number analyzed (Participants) | 129
  Change from Baseline at Week 168 [OD] | -0.004 (0.338)
  Change from Baseline at Week 168 [OS]: number analyzed (Participants) | 128
  Change from Baseline at Week 168 [OS] | -0.053 (0.324)
  Change from Baseline at Week 192 [OD]: number analyzed (Participants) | 131
  Change from Baseline at Week 192 [OD] | 0.008 (0.383)
  Change from Baseline at Week 192 [OS]: number analyzed (Participants) | 130
  Change from Baseline at Week 192 [OS] | -0.056 (0.386)
  Change from Baseline at Week 216 [OD]: number analyzed (Participants) | 124
  Change from Baseline at Week 216 [OD] | 0.019 (0.427)
  Change from Baseline at Week 216 [OS]: number analyzed (Participants) | 125
  Change from Baseline at Week 216 [OS] | -0.069 (0.440)
  Change from Baseline at Week 240 [OD]: number analyzed (Participants) | 117
  Change from Baseline at Week 240 [OD] | 0.007 (0.465)
  Change from Baseline at Week 240 [OS]: number analyzed (Participants) | 117
  Change from Baseline at Week 240 [OS] | -0.085 (0.490)
  Change from Baseline at Week 264 [OD]: number analyzed (Participants) | 118
  Change from Baseline at Week 264 [OD] | -0.016 (0.421)
  Change from Baseline at Week 264 [OS]: number analyzed (Participants) | 119
  Change from Baseline at Week 264 [OS] | -0.074 (0.472)
  Change from Baseline at Week 288 [OD]: number analyzed (Participants) | 109
  Change from Baseline at Week 288 [OD] | 0.006 (0.386)
  Change from Baseline at Week 288 [OS]: number analyzed (Participants) | 110
  Change from Baseline at Week 288 [OS] | -0.085 (0.458)
  Change from Baseline at Week 312 [OD]: number analyzed (Participants) | 98
  Change from Baseline at Week 312 [OD] | -0.043 (0.420)
  Change from Baseline at Week 312 [OS]: number analyzed (Participants) | 99
  Change from Baseline at Week 312 [OS] | -0.106 (0.499)
  Change from Baseline at Week 336 [OD]: number analyzed (Participants) | 92
  Change from Baseline at Week 336 [OD] | -0.025 (0.470)
  Change from Baseline at Week 336 [OS]: number analyzed (Participants) | 91
  Change from Baseline at Week 336 [OS] | -0.112 (0.539)
  Change from Baseline at Week 360 [OD]: number analyzed (Participants) | 87
  Change from Baseline at Week 360 [OD] | -0.008 (0.400)
  Change from Baseline at Week 360 [OS]: number analyzed (Participants) | 86
  Change from Baseline at Week 360 [OS] | -0.122 (0.524)
  Change from Baseline at Week 384 [OD]: number analyzed (Participants) | 72
  Change from Baseline at Week 384 [OD] | 0.002 (0.421)
  Change from Baseline at Week 384 [OS]: number analyzed (Participants) | 71
  Change from Baseline at Week 384 [OS] | -0.086 (0.467)
  Change from Baseline at Week 408 [OD]: number analyzed (Participants) | 55
  Change from Baseline at Week 408 [OD] | 0.039 (0.466)
  Change from Baseline at Week 408 [OS]: number analyzed (Participants) | 54
  Change from Baseline at Week 408 [OS] | -0.071 (0.572)
  Change from Baseline at Week 432 [OD]: number analyzed (Participants) | 50
  Change from Baseline at Week 432 [OD] | -0.010 (0.427)
  Change from Baseline at Week 432 [OS]: number analyzed (Participants) | 49
  Change from Baseline at Week 432 [OS] | -0.145 (0.509)
  Change from Baseline at Week 456 [OD]: number analyzed (Participants) | 38
  Change from Baseline at Week 456 [OD] | 0.011 (0.373)
  Change from Baseline at Week 456 [OS]: number analyzed (Participants) | 38
  Change from Baseline at Week 456 [OS] | -0.109 (0.509)
  Change from Baseline at Week 480 [OD]: number analyzed (Participants) | 18
  Change from Baseline at Week 480 [OD] | -0.106 (0.315)
  Change from Baseline at Week 480 [OS]: number analyzed (Participants) | 17
  Change from Baseline at Week 480 [OS] | -0.018 (0.185)
  Change from Baseline at Week 504 [OD]: number analyzed (Participants) | 2
  Change from Baseline at Week 504 [OD] | -0.200 (0.141)
  Change from Baseline at Week 504 [OS]: number analyzed (Participants) | 2
  Change from Baseline at Week 504 [OS] | -0.320 (0.283)
  Change from Baseline at Week 528 [OD]: number analyzed (Participants) | 1
  Change from Baseline at Week 528 [OD] | 0.220 (NA) — Since only 1 participant was analyzed, SD could not be calculated.
  Change from Baseline at Week 528 [OS]: number analyzed (Participants) | 1
  Change from Baseline at Week 528 [OS] | 0.300 (NA) — Since only 1 participant was analyzed, SD could not be calculated.

14. Secondary Outcome: Concentrations of Interleukin-6 (IL-6) in Blood
Description: Baseline was defined as last observation collected on or before day of first study drug administration in parent studies (NCT02028884/NCT02073279). All data from the time of randomization in the parent studies up to the end of study WN42349 for satralizumab-treated participants are reported here.
Time Frame: Baseline, every two weeks from Weeks 2 to 8; every 4 weeks from Weeks 12 to 192; every 24 weeks from Weeks 216 to 528
Population: All Participants-treated population included participants who received at least one dose of satralizumab at any time either during the parent studies or this study, irrespective of enrollment in current study. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms/millilitre (pg/mL)
Arm/Group | Satralizumab
Number analyzed (Participants) | 163
picograms/millilitre (pg/mL)
  Baseline | 2.07 (70.3)
  Week 2: number analyzed (Participants) | 101
  Week 2 | 21.27 (97.0)
  Week 4 | 21.90 (108.2)
  Week 8: number analyzed (Participants) | 159
  Week 8 | 19.35 (110.2)
  Week 12: number analyzed (Participants) | 157
  Week 12 | 18.84 (99.9)
  Week 16: number analyzed (Participants) | 151
  Week 16 | 17.53 (108.5)
  Week 20: number analyzed (Participants) | 157
  Week 20 | 17.16 (108.1)
  Week 24: number analyzed (Participants) | 152
  Week 24 | 17.77 (101.9)
  Week 28: number analyzed (Participants) | 152
  Week 28 | 17.08 (109.6)
  Week 32: number analyzed (Participants) | 151
  Week 32 | 18.32 (107.1)
  Week 36: number analyzed (Participants) | 145
  Week 36 | 18.29 (95.7)
  Week 40: number analyzed (Participants) | 141
  Week 40 | 16.21 (95.8)
  Week 44: number analyzed (Participants) | 145
  Week 44 | 17.59 (108.5)
  Week 48: number analyzed (Participants) | 141
  Week 48 | 18.59 (105.5)
  Week 52: number analyzed (Participants) | 93
  Week 52 | 18.55 (101.8)
  Week 56: number analyzed (Participants) | 91
  Week 56 | 18.78 (124.2)
  Week 60: number analyzed (Participants) | 90
  Week 60 | 20.56 (99.8)
  Week 64: number analyzed (Participants) | 87
  Week 64 | 20.04 (98.2)
  Week 68: number analyzed (Participants) | 83
  Week 68 | 19.70 (95.6)
  Week 72: number analyzed (Participants) | 83
  Week 72 | 18.48 (103.7)
  Week 76: number analyzed (Participants) | 80
  Week 76 | 18.05 (89.0)
  Week 80: number analyzed (Participants) | 71
  Week 80 | 17.93 (101.2)
  Week 84: number analyzed (Participants) | 74
  Week 84 | 18.44 (111.1)
  Week 88: number analyzed (Participants) | 69
  Week 88 | 20.33 (89.1)
  Week 92: number analyzed (Participants) | 68
  Week 92 | 17.12 (100.7)
  Week 96: number analyzed (Participants) | 69
  Week 96 | 19.72 (107.8)
  Week 100: number analyzed (Participants) | 63
  Week 100 | 19.73 (111.5)
  Week 104: number analyzed (Participants) | 66
  Week 104 | 19.34 (82.6)
  Week 108: number analyzed (Participants) | 66
  Week 108 | 19.74 (94.9)
  Week 112: number analyzed (Participants) | 65
  Week 112 | 21.39 (95.8)
  Week 116: number analyzed (Participants) | 60
  Week 116 | 17.98 (93.4)
  Week 120: number analyzed (Participants) | 60
  Week 120 | 19.26 (108.0)
  Week 124: number analyzed (Participants) | 60
  Week 124 | 18.41 (98.5)
  Week 128: number analyzed (Participants) | 59
  Week 128 | 18.17 (93.3)
  Week 132: number analyzed (Participants) | 59
  Week 132 | 17.83 (98.6)
  Week 136: number analyzed (Participants) | 53
  Week 136 | 19.22 (100.4)
  Week 140: number analyzed (Participants) | 51
  Week 140 | 17.62 (91.5)
  Week 144: number analyzed (Participants) | 62
  Week 144 | 16.54 (101.1)
  Week 148: number analyzed (Participants) | 50
  Week 148 | 18.95 (82.9)
  Week 152: number analyzed (Participants) | 44
  Week 152 | 19.71 (100.3)
  Week 156: number analyzed (Participants) | 37
  Week 156 | 20.84 (78.5)
  Week 160: number analyzed (Participants) | 43
  Week 160 | 19.91 (81.3)
  Week 164: number analyzed (Participants) | 38
  Week 164 | 19.76 (76.8)
  Week 168: number analyzed (Participants) | 54
  Week 168 | 22.33 (87.4)
  Week 172: number analyzed (Participants) | 34
  Week 172 | 21.94 (82.8)
  Week 176: number analyzed (Participants) | 32
  Week 176 | 23.31 (75.8)
  Week 180: number analyzed (Participants) | 35
  Week 180 | 21.28 (78.4)
  Week 184: number analyzed (Participants) | 29
  Week 184 | 23.23 (98.0)
  Week 188: number analyzed (Participants) | 35
  Week 188 | 23.52 (86.0)
  Week 192: number analyzed (Participants) | 62
  Week 192 | 22.25 (76.4)
  Week 216: number analyzed (Participants) | 62
  Week 216 | 19.41 (102.0)
  Week 240: number analyzed (Participants) | 66
  Week 240 | 18.22 (101.8)
  Week 264: number analyzed (Participants) | 61
  Week 264 | 18.56 (99.6)
  Week 288: number analyzed (Participants) | 67
  Week 288 | 19.17 (94.4)
  Week 312: number analyzed (Participants) | 68
  Week 312 | 21.70 (82.1)
  Week 336: number analyzed (Participants) | 85
  Week 336 | 17.71 (103.0)
  Week 360: number analyzed (Participants) | 86
  Week 360 | 19.40 (77.1)
  Week 384: number analyzed (Participants) | 68
  Week 384 | 19.68 (91.2)
  Week 408: number analyzed (Participants) | 56
  Week 408 | 18.94 (113.3)
  Week 432: number analyzed (Participants) | 50
  Week 432 | 19.29 (124.0)
  Week 456: number analyzed (Participants) | 36
  Week 456 | 17.90 (94.5)
  Week 480: number analyzed (Participants) | 18
  Week 480 | 20.89 (42.5)
  Week 504: number analyzed (Participants) | 2
  Week 504 | 8.40 (32.4)
  Week 528: number analyzed (Participants) | 1
  Week 528 | 13.50 (NA) — Since only 1 participant was analyzed, geometric coefficient of variation could not be calculated.

15. Secondary Outcome: Concentrations of Soluble IL-6 Receptor (sIL-6R) in Blood
Description: as for outcome 14
Time Frame: Baseline, every two weeks from Weeks 2 to 8; every 4 weeks from Weeks 12 to 192; every 24 weeks from Weeks 216 to 528
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/millilitre (ng/mL)
Arm/Group | Satralizumab
Number analyzed (Participants) | 164
nanograms/millilitre (ng/mL)
  Baseline | 32.27 (29.0)
  Week 2: number analyzed (Participants) | 102
  Week 2 | 404.20 (22.1)
  Week 4: number analyzed (Participants) | 163
  Week 4 | 536.46 (28.3)
  Week 8: number analyzed (Participants) | 161
  Week 8 | 566.91 (49.4)
  Week 12: number analyzed (Participants) | 159
  Week 12 | 568.96 (53.8)
  Week 16: number analyzed (Participants) | 152
  Week 16 | 561.69 (56.2)
  Week 20: number analyzed (Participants) | 157
  Week 20 | 543.99 (63.3)
  Week 24: number analyzed (Participants) | 154
  Week 24 | 556.84 (60.5)
  Week 28: number analyzed (Participants) | 154
  Week 28 | 547.77 (64.0)
  Week 32: number analyzed (Participants) | 153
  Week 32 | 574.72 (50.9)
  Week 36: number analyzed (Participants) | 146
  Week 36 | 552.54 (61.9)
  Week 40: number analyzed (Participants) | 142
  Week 40 | 556.08 (62.9)
  Week 44: number analyzed (Participants) | 150
  Week 44 | 569.26 (62.3)
  Week 48: number analyzed (Participants) | 143
  Week 48 | 575.25 (58.8)
  Week 52: number analyzed (Participants) | 93
  Week 52 | 555.92 (60.3)
  Week 56: number analyzed (Participants) | 93
  Week 56 | 523.80 (71.6)
  Week 60: number analyzed (Participants) | 91
  Week 60 | 549.23 (58.7)
  Week 64: number analyzed (Participants) | 88
  Week 64 | 550.61 (62.7)
  Week 68: number analyzed (Participants) | 83
  Week 68 | 581.62 (61.5)
  Week 72: number analyzed (Participants) | 84
  Week 72 | 540.99 (66.6)
  Week 76: number analyzed (Participants) | 81
  Week 76 | 519.20 (74.5)
  Week 80: number analyzed (Participants) | 71
  Week 80 | 535.83 (73.9)
  Week 84: number analyzed (Participants) | 74
  Week 84 | 533.47 (66.9)
  Week 88: number analyzed (Participants) | 69
  Week 88 | 523.64 (69.8)
  Week 92: number analyzed (Participants) | 70
  Week 92 | 515.37 (74.5)
  Week 96: number analyzed (Participants) | 70
  Week 96 | 526.59 (70.4)
  Week 100: number analyzed (Participants) | 64
  Week 100 | 534.72 (71.2)
  Week 104: number analyzed (Participants) | 66
  Week 104 | 583.53 (55.1)
  Week 108: number analyzed (Participants) | 66
  Week 108 | 578.63 (57.1)
  Week 112: number analyzed (Participants) | 65
  Week 112 | 594.60 (61.0)
  Week 116: number analyzed (Participants) | 60
  Week 116 | 571.37 (62.0)
  Week 120: number analyzed (Participants) | 61
  Week 120 | 615.02 (42.7)
  Week 124: number analyzed (Participants) | 61
  Week 124 | 590.17 (53.3)
  Week 128: number analyzed (Participants) | 60
  Week 128 | 559.85 (58.7)
  Week 132: number analyzed (Participants) | 59
  Week 132 | 580.53 (45.0)
  Week 136: number analyzed (Participants) | 55
  Week 136 | 607.27 (38.6)
  Week 140: number analyzed (Participants) | 52
  Week 140 | 592.84 (43.8)
  Week 144: number analyzed (Participants) | 62
  Week 144 | 571.70 (61.2)
  Week 148: number analyzed (Participants) | 50
  Week 148 | 610.47 (43.8)
  Week 152: number analyzed (Participants) | 44
  Week 152 | 565.34 (73.3)
  Week 156: number analyzed (Participants) | 38
  Week 156 | 667.59 (22.3)
  Week 160: number analyzed (Participants) | 43
  Week 160 | 652.90 (28.8)
  Week 164: number analyzed (Participants) | 38
  Week 164 | 636.27 (34.9)
  Week 168: number analyzed (Participants) | 54
  Week 168 | 662.43 (29.9)
  Week 172: number analyzed (Participants) | 34
  Week 172 | 643.84 (36.8)
  Week 176: number analyzed (Participants) | 32
  Week 176 | 670.38 (28.3)
  Week 180: number analyzed (Participants) | 35
  Week 180 | 655.31 (35.0)
  Week 184: number analyzed (Participants) | 30
  Week 184 | 684.07 (18.5)
  Week 188: number analyzed (Participants) | 35
  Week 188 | 666.52 (30.8)
  Week 192: number analyzed (Participants) | 62
  Week 192 | 611.46 (67.0)
  Week 216: number analyzed (Participants) | 63
  Week 216 | 592.12 (68.9)
  Week 240: number analyzed (Participants) | 71
  Week 240 | 587.26 (58.7)
  Week 264: number analyzed (Participants) | 63
  Week 264 | 570.35 (45.3)
  Week 288: number analyzed (Participants) | 67
  Week 288 | 572.20 (52.2)
  Week 312: number analyzed (Participants) | 68
  Week 312 | 608.11 (35.0)
  Week 336: number analyzed (Participants) | 85
  Week 336 | 533.73 (71.8)
  Week 360: number analyzed (Participants) | 87
  Week 360 | 557.05 (55.3)
  Week 384: number analyzed (Participants) | 69
  Week 384 | 549.57 (58.0)
  Week 408: number analyzed (Participants) | 56
  Week 408 | 586.95 (62.4)
  Week 432: number analyzed (Participants) | 50
  Week 432 | 569.09 (42.7)
  Week 456: number analyzed (Participants) | 36
  Week 456 | 561.16 (56.8)
  Week 480: number analyzed (Participants) | 18
  Week 480 | 652.16 (18.0)
  Week 504: number analyzed (Participants) | 2
  Week 504 | 668.04 (13.4)
  Week 528: number analyzed (Participants) | 1
  Week 528 | 910.00 (NA) — Since only 1 participant was analyzed, geometric coefficient of variation could not be calculated.

16. Secondary Outcome: Concentration of C-Reactive Protein (CRP) in Blood
Description: as for outcome 14
Time Frame: Baseline, every two weeks from Weeks 2 to 8; every 4 weeks from Weeks 12 to 192; every 24 weeks from Weeks 216 to 528
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams/litre (mg/L)
Arm/Group | Satralizumab
Number analyzed (Participants) | 165
milligrams/litre (mg/L)
  Baseline | 1.27 (226.6)
  Week 2: number analyzed (Participants) | 102
  Week 2 | 0.38 (118.0)
  Week 4: number analyzed (Participants) | 162
  Week 4 | 0.36 (113.3)
  Week 8: number analyzed (Participants) | 161
  Week 8 | 0.39 (125.9)
  Week 12: number analyzed (Participants) | 156
  Week 12 | 0.42 (144.9)
  Week 16: number analyzed (Participants) | 152
  Week 16 | 0.42 (151.1)
  Week 20: number analyzed (Participants) | 157
  Week 20 | 0.41 (157.8)
  Week 24: number analyzed (Participants) | 154
  Week 24 | 0.44 (161.0)
  Week 28: number analyzed (Participants) | 155
  Week 28 | 0.41 (175.7)
  Week 32: number analyzed (Participants) | 153
  Week 32 | 0.44 (171.4)
  Week 36: number analyzed (Participants) | 147
  Week 36 | 0.43 (185.3)
  Week 40: number analyzed (Participants) | 146
  Week 40 | 0.48 (184.3)
  Week 44: number analyzed (Participants) | 150
  Week 44 | 0.43 (182.3)
  Week 48: number analyzed (Participants) | 144
  Week 48 | 0.44 (167.9)
  Week 52: number analyzed (Participants) | 91
  Week 52 | 0.50 (177.4)
  Week 56: number analyzed (Participants) | 91
  Week 56 | 0.47 (183.8)
  Week 60: number analyzed (Participants) | 91
  Week 60 | 0.49 (183.3)
  Week 64: number analyzed (Participants) | 88
  Week 64 | 0.47 (177.6)
  Week 68: number analyzed (Participants) | 85
  Week 68 | 0.52 (194.3)
  Week 72: number analyzed (Participants) | 89
  Week 72 | 0.50 (223.7)
  Week 76: number analyzed (Participants) | 81
  Week 76 | 0.51 (189.5)
  Week 80: number analyzed (Participants) | 72
  Week 80 | 0.51 (200.4)
  Week 84: number analyzed (Participants) | 74
  Week 84 | 0.53 (227.4)
  Week 88: number analyzed (Participants) | 69
  Week 88 | 0.51 (188.0)
  Week 92: number analyzed (Participants) | 69
  Week 92 | 0.51 (200.4)
  Week 96: number analyzed (Participants) | 71
  Week 96 | 0.52 (183.4)
  Week 100: number analyzed (Participants) | 64
  Week 100 | 0.52 (231.4)
  Week 104: number analyzed (Participants) | 66
  Week 104 | 0.46 (167.3)
  Week 108: number analyzed (Participants) | 66
  Week 108 | 0.51 (161.9)
  Week 112: number analyzed (Participants) | 66
  Week 112 | 0.48 (191.7)
  Week 116: number analyzed (Participants) | 61
  Week 116 | 0.43 (177.0)
  Week 120: number analyzed (Participants) | 64
  Week 120 | 0.52 (227.6)
  Week 124: number analyzed (Participants) | 61
  Week 124 | 0.56 (173.2)
  Week 128: number analyzed (Participants) | 60
  Week 128 | 0.57 (209.1)
  Week 132: number analyzed (Participants) | 61
  Week 132 | 0.59 (234.8)
  Week 136: number analyzed (Participants) | 59
  Week 136 | 0.54 (193.9)
  Week 140: number analyzed (Participants) | 55
  Week 140 | 0.61 (283.9)
  Week 144: number analyzed (Participants) | 65
  Week 144 | 0.47 (205.6)
  Week 148: number analyzed (Participants) | 51
  Week 148 | 0.47 (152.0)
  Week 152: number analyzed (Participants) | 46
  Week 152 | 0.51 (147.8)
  Week 156: number analyzed (Participants) | 43
  Week 156 | 0.47 (129.5)
  Week 160: number analyzed (Participants) | 45
  Week 160 | 0.48 (148.9)
  Week 164: number analyzed (Participants) | 39
  Week 164 | 0.49 (163.7)
  Week 168: number analyzed (Participants) | 56
  Week 168 | 0.45 (148.9)
  Week 172: number analyzed (Participants) | 32
  Week 172 | 0.45 (228.2)
  Week 176: number analyzed (Participants) | 33
  Week 176 | 0.39 (156.7)
  Week 180: number analyzed (Participants) | 35
  Week 180 | 0.42 (156.6)
  Week 184: number analyzed (Participants) | 33
  Week 184 | 0.38 (197.3)
  Week 188: number analyzed (Participants) | 37
  Week 188 | 0.46 (154.0)
  Week 192: number analyzed (Participants) | 71
  Week 192 | 0.40 (188.5)
  Week 216: number analyzed (Participants) | 62
  Week 216 | 0.30 (110.4)
  Week 240: number analyzed (Participants) | 78
  Week 240 | 0.40 (221.9)
  Week 264: number analyzed (Participants) | 65
  Week 264 | 0.36 (178.6)
  Week 288: number analyzed (Participants) | 68
  Week 288 | 0.36 (215.6)
  Week 312: number analyzed (Participants) | 68
  Week 312 | 0.32 (160.2)
  Week 336: number analyzed (Participants) | 84
  Week 336 | 0.48 (302.7)
  Week 360: number analyzed (Participants) | 89
  Week 360 | 0.39 (221.2)
  Week 384: number analyzed (Participants) | 74
  Week 384 | 0.37 (185.9)
  Week 408: number analyzed (Participants) | 56
  Week 408 | 0.29 (195.5)
  Week 432: number analyzed (Participants) | 51
  Week 432 | 0.35 (161.1)
  Week 456: number analyzed (Participants) | 39
  Week 456 | 0.32 (139.8)
  Week 480: number analyzed (Participants) | 21
  Week 480 | 0.17 (33.0)
  Week 504: number analyzed (Participants) | 3
  Week 504 | 0.15 (0.0)
  Week 528: number analyzed (Participants) | 1
  Week 528 | 0.15 (NA) — Since only 1 participant was analyzed, geometric coefficient of variation could not be calculated.

17. Secondary Outcome: Serum Concentration of Satralizumab at Specified Timepoints
Description: as for outcome 14
Time Frame: Baseline, Week 2, Week 4, Week 5, Week 6; every 4 weeks from Weeks 8 to 192; every 24 weeks from Weeks 216 to 528
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/litre (ng/L)
Arm/Group | Satralizumab
Number analyzed (Participants) | 164
nanograms/litre (ng/L)
  Baseline | 103.75 (29.7)
  Week 2: number analyzed (Participants) | 102
  Week 2 | 7489.76 (102.8)
  Week 4: number analyzed (Participants) | 155
  Week 4 | 14631.06 (95.9)
  Week 5: number analyzed (Participants) | 64
  Week 5 | 20068.86 (105.6)
  Week 6: number analyzed (Participants) | 62
  Week 6 | 17495.09 (157.7)
  Week 8: number analyzed (Participants) | 160
  Week 8 | 12673.14 (190.9)
  Week 12: number analyzed (Participants) | 158
  Week 12 | 11031.23 (220.8)
  Week 16: number analyzed (Participants) | 152
  Week 16 | 10588.85 (250.6)
  Week 20: number analyzed (Participants) | 157
  Week 20 | 10065.62 (305.1)
  Week 24: number analyzed (Participants) | 154
  Week 24 | 10605.69 (306.1)
  Week 28: number analyzed (Participants) | 154
  Week 28 | 9730.68 (333.9)
  Week 32: number analyzed (Participants) | 153
  Week 32 | 10686.86 (282.5)
  Week 36: number analyzed (Participants) | 146
  Week 36 | 10036.31 (368.4)
  Week 40: number analyzed (Participants) | 143
  Week 40 | 9508.64 (400.1)
  Week 44: number analyzed (Participants) | 150
  Week 44 | 9891.10 (361.9)
  Week 48: number analyzed (Participants) | 144
  Week 48 | 11282.31 (311.3)
  Week 52: number analyzed (Participants) | 93
  Week 52 | 9585.58 (500.8)
  Week 56: number analyzed (Participants) | 93
  Week 56 | 9209.84 (468.2)
  Week 60: number analyzed (Participants) | 91
  Week 60 | 10090.62 (394.0)
  Week 64: number analyzed (Participants) | 88
  Week 64 | 9186.35 (376.7)
  Week 68: number analyzed (Participants) | 83
  Week 68 | 9951.51 (359.5)
  Week 72: number analyzed (Participants) | 131
  Week 72 | 10737.11 (340.8)
  Week 76: number analyzed (Participants) | 82
  Week 76 | 8414.98 (522.7)
  Week 80: number analyzed (Participants) | 74
  Week 80 | 8557.82 (431.6)
  Week 84: number analyzed (Participants) | 77
  Week 84 | 8208.84 (473.6)
  Week 88: number analyzed (Participants) | 73
  Week 88 | 8457.80 (498.3)
  Week 92: number analyzed (Participants) | 71
  Week 92 | 8316.17 (510.7)
  Week 96: number analyzed (Participants) | 119
  Week 96 | 10560.87 (329.6)
  Week 100: number analyzed (Participants) | 70
  Week 100 | 9841.13 (361.2)
  Week 104: number analyzed (Participants) | 68
  Week 104 | 11256.29 (278.2)
  Week 108: number analyzed (Participants) | 71
  Week 108 | 10521.75 (273.5)
  Week 112: number analyzed (Participants) | 71
  Week 112 | 10362.73 (314.0)
  Week 116: number analyzed (Participants) | 63
  Week 116 | 11219.11 (331.1)
  Week 120: number analyzed (Participants) | 105
  Week 120 | 11619.05 (315.4)
  Week 124: number analyzed (Participants) | 66
  Week 124 | 9680.42 (354.6)
  Week 128: number analyzed (Participants) | 62
  Week 128 | 8727.98 (362.3)
  Week 132: number analyzed (Participants) | 65
  Week 132 | 8378.76 (437.7)
  Week 136: number analyzed (Participants) | 61
  Week 136 | 10182.79 (294.2)
  Week 140: number analyzed (Participants) | 57
  Week 140 | 9731.57 (440.3)
  Week 144: number analyzed (Participants) | 101
  Week 144 | 11206.52 (328.4)
  Week 148: number analyzed (Participants) | 56
  Week 148 | 11605.26 (291.6)
  Week 152: number analyzed (Participants) | 45
  Week 152 | 12065.91 (352.8)
  Week 156: number analyzed (Participants) | 45
  Week 156 | 13017.85 (222.9)
  Week 160: number analyzed (Participants) | 50
  Week 160 | 13952.43 (173.1)
  Week 164: number analyzed (Participants) | 43
  Week 164 | 13869.87 (202.0)
  Week 168: number analyzed (Participants) | 85
  Week 168 | 14256.36 (183.0)
  Week 172: number analyzed (Participants) | 42
  Week 172 | 13018.63 (227.2)
  Week 176: number analyzed (Participants) | 37
  Week 176 | 11989.36 (330.9)
  Week 180: number analyzed (Participants) | 42
  Week 180 | 15333.00 (150.7)
  Week 184: number analyzed (Participants) | 43
  Week 184 | 16449.28 (101.1)
  Week 188: number analyzed (Participants) | 43
  Week 188 | 14519.13 (221.7)
  Week 192: number analyzed (Participants) | 106
  Week 192 | 11926.93 (284.9)
  Week 216: number analyzed (Participants) | 123
  Week 216 | 10582.11 (404.7)
  Week 240: number analyzed (Participants) | 114
  Week 240 | 13683.03 (237.7)
  Week 264: number analyzed (Participants) | 116
  Week 264 | 11576.23 (326.0)
  Week 288: number analyzed (Participants) | 108
  Week 288 | 13169.85 (221.9)
  Week 312: number analyzed (Participants) | 96
  Week 312 | 13007.87 (243.1)
  Week 336: number analyzed (Participants) | 91
  Week 336 | 10522.02 (407.6)
  Week 360: number analyzed (Participants) | 87
  Week 360 | 11604.67 (295.8)
  Week 384: number analyzed (Participants) | 70
  Week 384 | 14508.95 (303.3)
  Week 408: number analyzed (Participants) | 56
  Week 408 | 14652.75 (290.3)
  Week 432: number analyzed (Participants) | 49
  Week 432 | 13287.68 (329.1)
  Week 456: number analyzed (Participants) | 36
  Week 456 | 18532.35 (174.8)
  Week 480: number analyzed (Participants) | 19
  Week 480 | 26688.35 (56.3)
  Week 504: number analyzed (Participants) | 2
  Week 504 | 43917.08 (8.7)
  Week 528: number analyzed (Participants) | 1
  Week 528 | 57800.00 (NA) — Since only 1 participant was analyzed, geometric coefficient of variation could not be calculated.

18. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs) From the First Dose of Satralizumab in Studies NCT02028884 or NCT02073279
Description: The number and percentage of ADA-positive participants and ADA-negative participants at baseline (baseline prevalence) and after drug administration (post-baseline incidence) were summarized. Baseline evaluable participants were participants with an ADA assay result at baseline. Post-baseline evaluable participants were participants with an ADA assay from at least one post-baseline sample. Participants positive for ADA= number of participants with positive ADA result. Participants negative for ADA=number of participants with negative or missing baseline ADA result(s) and all negative post-baseline results. Baseline was defined as last observation collected on or before day of first study drug administration in parent studies. All data from the time of randomization in the parent studies up to the end of study WN42349 for satralizumab-treated participants are reported here.
Time Frame: First dose of satralizumab in parent studies up to end of study WN42349 (up to 523 weeks)
Population: All Participants-treated population included participants who received at least one dose of satralizumab at any time either during the parent studies or this study, irrespective of enrollment in current study. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Satralizumab
Number analyzed (Participants) | 166
Participants
  Baseline: number analyzed (Participants) | 164
  Baseline: Positive | 3
  Baseline: Negative | 161
  Post-baseline: Positive | 99
  Post-baseline: Negative | 67

ADVERSE EVENTS:
Time Frame: Baseline up to 523 weeks
Description: All Participants-treated population included participants who received at least one dose of satralizumab at any time either during the parent studies or this study. Participants from parent studies who did not enroll in the current study but received at least one dose satralizumab are also considered in this analysis set. The first dosing visit in the current study or the first satralizumab dosing visit in the parent studies (NCT02028884/NCT02073279) was considered as baseline for this study.
Arm/Group | Satralizumab
All-Cause Mortality (participants affected / at risk) | 0/166
Serious Adverse Events (participants affected / at risk) | 44/166
Other Adverse Events (participants affected / at risk) | 155/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Satralizumab (N=166)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Hypothermia (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Atypical mycobacterial infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 2 (3)
Hepatitis E (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 3 (3)
Large intestine infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5)
Pulmonary sepsis (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Septic endocarditis (Infections and infestations) | 1 (1)
Sinusitis fungal (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Urosepsis (Infections and infestations) | 2 (2)
Accidental exposure to product (Injury, poisoning and procedural complications) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (2)
Fracture displacement (Injury, poisoning and procedural complications) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1)
Limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Migraine (Nervous system disorders) | 1 (1)
Neuromyelitis optica pseudo relapse (Nervous system disorders) | 1 (1)
Parkinsonism (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (2)
Tension headache (Nervous system disorders) | 1 (1)
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2)
Suicide attempt (Psychiatric disorders) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 2 (2)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rehabilitation therapy (Surgical and medical procedures) | 1 (1)
Aneurysm (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Satralizumab (N=166)
Anaemia (Blood and lymphatic system disorders) | 15 (19)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 9 (12)
Leukopenia (Blood and lymphatic system disorders) | 18 (33)
Lymphopenia (Blood and lymphatic system disorders) | 10 (27)
Neutropenia (Blood and lymphatic system disorders) | 16 (26)
Abdominal pain upper (Gastrointestinal disorders) | 11 (12)
Constipation (Gastrointestinal disorders) | 18 (23)
Dental caries (Gastrointestinal disorders) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 21 (42)
Nausea (Gastrointestinal disorders) | 21 (27)
Toothache (Gastrointestinal disorders) | 11 (14)
Vomiting (Gastrointestinal disorders) | 9 (11)
Fatigue (General disorders) | 17 (22)
Oedema peripheral (General disorders) | 11 (13)
COVID-19 (Infections and infestations) | 31 (33)
Cystitis (Infections and infestations) | 15 (18)
Ear infection (Infections and infestations) | 10 (13)
Gastroenteritis (Infections and infestations) | 9 (17)
Influenza (Infections and infestations) | 13 (14)
Nasopharyngitis (Infections and infestations) | 48 (132)
Oral herpes (Infections and infestations) | 9 (70)
Sinusitis (Infections and infestations) | 16 (22)
Upper respiratory tract infection (Infections and infestations) | 46 (172)
Urinary tract infection (Infections and infestations) | 40 (139)
Fall (Injury, poisoning and procedural complications) | 11 (21)
Injection related reaction (Injury, poisoning and procedural complications) | 24 (57)
Ligament sprain (Injury, poisoning and procedural complications) | 9 (11)
Alanine aminotransferase increased (Investigations) | 14 (20)
Blood cholesterol increased (Investigations) | 14 (23)
Blood creatine phosphokinase increased (Investigations) | 10 (12)
Blood fibrinogen decreased (Investigations) | 10 (17)
Complement factor C4 decreased (Investigations) | 9 (11)
Lymphocyte count decreased (Investigations) | 11 (17)
White blood cell count decreased (Investigations) | 13 (30)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 9 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 35 (43)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (31)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 (43)
Dizziness (Nervous system disorders) | 15 (20)
Headache (Nervous system disorders) | 44 (86)
Hypoaesthesia (Nervous system disorders) | 15 (24)
Anxiety (Psychiatric disorders) | 10 (11)
Depression (Psychiatric disorders) | 11 (14)
Insomnia (Psychiatric disorders) | 17 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (22)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 17 (21)
Eczema (Skin and subcutaneous tissue disorders) | 10 (11)
Rash (Skin and subcutaneous tissue disorders) | 20 (27)
Hypertension (Vascular disorders) | 11 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT04660539/Prot_SAP_000.pdf